CLINICAL TRIAL: NCT03448341
Title: Clinical and Instrumental Evaluation of Late Dysphagia in Naso and Oropharynx Cancer After Swallowing-organs (SWOARs)-Sparing Chemo-IMRT
Brief Title: Dysphagia Assessment After Swallowing Sparing RadioTherapy
Acronym: DASRT
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Stefano Ursino, MD, Researcher, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: 1112
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Cancer of Oropharynx; Cancer of Nasopharynx
Keywords: Radiotherapy; IMRT; Dysphagia; Oropharynx; Nasopharynx; FEES; VFS; Chemotherapy
MeSH Terms: conditions — Oropharyngeal Neoplasms; Nasopharyngeal Neoplasms; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To prospectively assess post-radiation late dysphagia by using MDADI questionnaire (deglutition-related quality of life) and objective instrumental assessment by means of Fiberoptic Endoscopic Evaluation of Swallowing (FEES) and Videofluoroscopy (VFS) in patients affected by nasopharynx and oropharynx cancers candidates to radiochemotherapy. Radiotherapy is delivered by using Intensity and Modulated Technique (IMRT) with a planning dose optimization to the swallowing related structures (SWOARs-sparing IMRT).

The primary aim is to assess the variations of MDADI, FEES and VFS from baseline to 6 and 12 months after treatment.

The secondary aim is to correlate clinical and instrumental results as well as radiation dose received by the different swallowing related structures (SWOARs) to the variations of clinical (MDADI) and instrumental (FEES and VFS) scores.

DETAILED DESCRIPTION:
The aim of the study is to prospectively investigate the impact of radiochemotherapy on both the deglution-related quality of life (QoL) by means of MDADI questionnaire and the swallowing function by means of Fiberoptic Endoscopic Evaluation of Swallowing (FEES) and Videofluoroscopy (VFS).

Radiotherapy All patients requiring bilateral neck irradiation will be considered.

The clinical target volumes (CTVs) is directly delineated by the radiation oncologist according to the guidelines of the Italian Association of Radiation Oncology-Head and Neck Working Group 27 and the corresponding planning target volumes (PTVs) is automatically created by uniform expansions of 0.3 cm.

Patients positioning is assessed by weekly cone beam CT (CBCT) and online correction to reduce systematic set-up errors.

The prescribed doses is 66 Gy at 2.2 Gy per fraction to the high risk gross volume PTV and 60-54 Gy at 2.0-1.8 Gy per fraction to the intermediate (optional) and low risk subclinical PTVs, respectively, delivered concomitantly in 30 daily fractions.

Eight different SWOARs are defined in each CT slice and included in IMRT planning objective functions: superior, middle and inferior constrictor muscle (SPCM, MPCM and IPCM), supraglottic larynx (SL), glottis larynx (GL), cricopharyngeus muscle (CPM) and cervical oesophagus (CE). Thereafter, the mean dose received by each swallowing structures as well as by parotid glands and oral cavity will be recorded.

In the IMRT optimisation cost function, target coverage replace sparing of any SWOARs, parotid glands and oral cavity, but the spinal cord.

The IMRT plans set target prescription goals and spinal cord maximum dose (Dmax) as the highest priority, whereas SWOAR constraints are set as secondary.

Medical therapy

Chemotherapy is given weekly using Cisplatin 40 mg/mq for a maximum of 6 cycles or 100 mg/mq every 3 weeks during the 6-week RT course for a maximum of 3 cycles.

MDADI questionnaire

All the enrolled patients fill in the MDADI questionnaire at baseline and at 6 and 12 months after ChemoRT. The validated Italian version of MDADI is used. A MDADI score of at least 80 represents an "optimal" deglutition-related QoL, a score between 60 and 80 represents an "adequate" deglutition-related QoL, and a score less than 60 represents a "poor" deglutition-related QoL. A 10-point difference in the MDADI composite score is considered a minimal clinically important difference (MCID) in the deglutition-related QoL.

Fiberoptic Endoscopic Evaluation of Swallowing (FEES)

This exam is specifically used to evaluate the severity of post-swallowing pharyngeal residue according to Farneti pooling score (P-score), a reliable and validated tool that significantly predicts aspirations.

Videofluoroscopy (VFS)

This exam is specifically used to evaluate the pattern of penetration and aspiration based on the Penetration-Aspiration Scale (PAS)

ELIGIBILITY:
Inclusion Criteria

1. Histological diagnosis of squamous cell carcinoma or undifferentiated carcinoma of the otoiatric district
2. Subsider of the primitive: (Nasopharynx Stage II and III); Oropharynx Stage III-IVA
3. ECOG Status 0-2
4. Chemiotherapy concomitant at radiotherapy (Cisplatin 100mg / m2 every 21 days or 40mg / m2 weekly)

Exclusion criteria

1. Histological diagnosis different from squamous or undifferentiated cell carcinoma
2. Subsider of the primitive different from Nasopharynx, Oropharynx
3. Nasopharynx Stage IV; Oropharynx Stage IVB and C
4. ECOG ≥3
5. Prior induction chemotherapy
6. Prior oncological surgery on the otoiatric district
7. Prior radiation treatment on the otoiatric district
8. Concomitant diseases that could modify the swallowing function (ex Amyotrophic Lateral Sclerosis or Multiple Sclerosis)
9. A history of excessive use of benzodiazepines or similar (ex patients in psychiatric therapy) or eostroesophageal reflux resistant at medical therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Locally Advanced Oropharynx or Nasopharynx cancer, that can be treated with an exclusive chemo-radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2016-07-16 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
To assess the changes of deglutition-related quality of life by means of MDADI questionnaire from before to after radiochemotherapy | Baseline, 6 and 12 months treatment
  All patients will be evaluated by using MDADI questionnaire at baseline and at 6 and 12 months after radiochemotherapy. The variations of MDADI questionnaire scores from before to after treatment will be analysed.
To assess the changes of deglutition function by means of Fiberoptic Endoscopic Evaluation of Swallowing (FEES) from before to after radiochemotherapy | Before, 6 and 12 months after treatment
  All patients will be evaluated by using FEES at baseline and at 6 and 12 months after radiochemotherapy. The variations of FEES scores from before to after treatment will be analysed
To assess the changes of deglutition function by means of Videofluoroscopy (VFS) from before to after radiochemotherapy | Before, 6 and 12 months after treatment
  All patients will be evaluated by using VFS at baseline and at 6 and 12 months after radiochemotherapy. The variations of VFS scores from before to after treatment will be analysed

SECONDARY OUTCOMES:
To correlate MDADI score (deglutition-related quality of life) changes with FEES and VFS score (deglutition function) changes from before to after treatment | Before, 6 and 12 months after treatment
  The correlation between clinical (MDADI) and instrumental (FEES and VFS) scores will be performed according to the following dichotomy:
  MDADI >80 vs MDADI <80 (optimal vs adequate or poor) FEES P-score 4-7 vs 8-11 (no/mild dysphagia vs adequate/severe dysphagia) VFS PAS score 1-2 vs 3-8 (safe deglutition vs penetration or aspiration)
To correlate radiation dose features received by the different swallowing related structures (SWOARs) to the changes of MDADI, FEES and VFS scores from before to after treatment by using a Machine Learning Methodology | At baseline and at 6 and 12 months
  Correlation between MDADI, FEES and VFS score changes with radiation dose received by the SWOARs will be performed according to the following criteria.
  The following radiation dose features (Gy) will be extracted for each SWOAR from dose volume hystograms (DVHs): V35, V45, V55, V65, minimum dose (Dmin), maximum dose (Dmax), mean dose (Dmean) and the dose corresponding to the absolute maximum of the differential DVH, hence the modal dose (Dmp).
  The abovementioned dose features will be correlated with the following outcome measures and according to the following stratification criteria:
  MDADI >80 vs MDADI <80 (optimal vs adequate or poor) FEES P-score 4-7 vs 8-11 (no/mild dysphagia vs adequate/severe dysphagia) VFS PAS score 1-2 vs 3-8 (safe deglutition vs penetration or aspiration)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Pisana, Pisa, Italy